CLINICAL TRIAL: NCT03289611
Title: Preeclampsia Ratio (sFlt-1/PlGF) Evaluation for Clinical and Obstetrical Guidance
Brief Title: Preeclampsia Ratio (sFlt-1/PlGF)
Acronym: PRECOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P161101
Record Dates: First submitted 2017-09-04; First posted 2017-09-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; pregnancy; biomarkers; prediction; safety; cost
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual management
- Experimental (Experimental): Ambulatory management if sFlt-1 / PlGF ratio is below 38 Usual management if sFlt-1/PlGF is between 38 and 85. If the ratio is > 85, monitoring will be intensified and patient hospitalization will be continued
  Interventions: Biological: sFlt-1 / PlGF ratio

INTERVENTIONS:
Biological: sFlt-1 / PlGF ratio — * Ambulatory management if sFlt-1 / PlGF ratio is below 38
  * usual management if sFlt-1/PlGF is between 38 and 85.
  * If the ratio is > 85, monitoring will be intensified and patient hospitalization will be continued
  Arms: Experimental

SUMMARY:
The aim of the PRECOG study is to determine in a prospective interventional randomized study whether the implementation of a predictive test based on the sFLT-1/PlGF ratio improves perinatal care and reduces costs, in patients with suspected preeclampsia before 35 weeks of gestation.

DETAILED DESCRIPTION:
Preeclampsia is a hypertensive disorder of pregnancy associated with placental insufficiency and is one of the major important of prematurity and maternal mortality worldwide. It complicates 2 to 7% of pregnancies. It is currently considered that preeclampsia is associated with maternal endothelial dysfunction induced by the release into the maternal circulation of excess placental factors (such as sFLT-1 a soluble receptor for VEGF and PlGF). There is currently no curative treatment, and only childbirth and delivery of the placenta alleviate the mother's symptoms. Moreover, the evolution from case with mild symptoms to a severe case of preeclampsia is often is often rapid and difficult to anticipate. Therefore, it is recommended to manage patients with preeclampsia in hospital and cases of suspected preeclampsia are usually admitted in prenatal units. Each year thousands of patients are hospitalized for surveillance and blood/urine analysis to rule out the diagnosis of preeclampsia. A biological test to predict preeclampsia would therefore be of particular interest in order to:

* identify patients without preeclampsia and therefore void costs and iatrogenic complications related to unnecessary hospitalization
* identify patients at high risk of maternal and perinatal complications in order to anticipate in utero transfer, optimize maternal and fetal surveillance and administrate steroids.

It has recently been demonstrated that sFLT-1 and PlGF have a high predictive value for the diagnosis and the prediction of preeclampsia, but the interest of introducing these markers in clinical practice has not been demonstrated yet. The diagnostic and predictive value of the sFlt-1/PlGF ratio in patients at risk of placenta-related disorders has been shown in the recent literature and estimation of the sFlt-1/PlGF ratio has become an additional tool in the management of these disorders, primarily PE. This ratio can distinguish the patients that develop maternal or perinatal complications in the next 7-14 days from those with uncomplicated pregnancy. Women with an sFlt-1/PlGF ratio<38 do not have PE at the time of the test and in all likelihood will not develop PE for at least 1week; it is thereby of great value for reassuring the clinician and the patient. Up to 80% of patients are supposed to be in this patient group; therefore, clinicians are able to exclude the majority of patients and focus on those who need more attention and care. On contrary women with a sFlt-1/PlGF ratio > 38 and more specifically those with a ratio over 85 are highly likely to develop preeclampsia and should be managed according to local practice/guidelines. Thus the use of such predictive tool appear very promising but its interest has not been demonstrated in prospective intervention studies.

The aim of the PRECOG study is to determine in a prospective interventional randomized study whether the implementation of a predictive test based on the sFLT-1/PlGF ratio improves perinatal care and reduces costs, in patients with suspected preeclampsia before 35 WG. costs, in patients with suspected preeclampsia before 35 WG.

ELIGIBILITY:
Inclusion Criteria:

Patient hospitalized for suspected preeclampsia between 24WG+ 0 days and 35WG + 6 days,

Patiente with at least one of the following criteria:

* Arterial hypertension defined by systolic BP ≥ 140 mm Hg or diastolic blood pressure ≥ 90 mm Hg
* Proteinuria greater than 0.3g / 24h or 0.3g / l or ≥ 3+
* Proteinuria / creatinine ratio ≥ 30 mg / mmol
* Pain in the epigastric bar
* Generalized edema
* Hepatic cytolysis> 1.5N
* Thrombocytopenia <150000 / mm3 Informed consent signed by both parties Non-opposition was accepted by parental authority Age ≥ 18 years

Exclusion Criteria:

Diagnosis of preeclampsia (arterial pressure> 140/90 and proteinuria> 0.3g / 24h or urine test> 3+) or complete HELLP syndrome (Platelets <100000 / mm3 and SGOT> 2N and LDH and collapsed Haptoglobin)

IUGR with absent or reverse diastolic umbilical flow

Fetal heart rate abnormalities

Gestational age <24 WG and> 35 WG

Multiple pregnancy

Patient without health insurance

Non-consent of patient

Minor patient

Congenital malformation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
number of patients hospitalised for more than 24 hours | up to 12 weeks
  Duration in hours, from admission to discharge from hospital at initial hospitalisation

SECONDARY OUTCOMES:
Maternal and fetal morbidity | up to 13 weeks
  severe preeclampsia, eclampsia, HELLP syndrome, Disseminated intravascular coagulation, abruptio placenta, delivery before 34 WA, IUGR< 3°P, Fetal death
Maternal morbidity | up to 13 weeks
  High blood pressure, preeclampsia, caesarean section, postpartum hemorrhage> 500 ml
Severe Maternal morbidity (Composite outcome ) | up to 13 weeks
  eclampsia, HELLP syndrome, Disseminated intravascular coagulation, Abruption placenta
Number of days between randomisation and delivery | up to 12 weeks
  Number of days between randomisation and delivery
Mode of delivery | At delivery
  Cesarean, vaginal delivery
Gestational age | at delivery
  Gestational age at delivery
Birth weight centile | At delivery
  Centile of birth weight
Fetal death | up to 13 weeks
  Fetal death diagnosed at ultrasound before delivery
Prematurity before 37 WG | up to 13 weeks
  Delivery before 37 WG + 0 days
Prematurity before 34 WG | Delivery
  Delivery before 34 WG + 0 days
Prematurity before 32 WG | Delivery
  Delivery before 32 WG + 0 days
Perinatal morbidity (Composite outcome) | At delivery
  prematurity, birth weight <10 ° P
Severe Perinatal morbidity (Composite outcome) | At delivery
  perinatal mortality, prematurity <34 SA, birth weight <3 ° P
Costs | up to 14 weeks
  direct costs of prenatal care, direct costs of neonatal care, total costs
Satisfaction form | Day 3 after delivery
  Satisfaction concerning the management of pregnancy and duration of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Jean GUIBOURDENCHE, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Cochin, Maternité Port Royal, Paris, France

REFERENCES:
- [Background] Tsatsaris V, Goffin F, Munaut C, Brichant JF, Pignon MR, Noel A, Schaaps JP, Cabrol D, Frankenne F, Foidart JM. Overexpression of the soluble vascular endothelial growth factor receptor in preeclamptic patients: pathophysiological consequences. J Clin Endocrinol Metab. 2003 Nov;88(11):5555-63. doi: 10.1210/jc.2003-030528. PMID 14602804
- [Background] Sibiude J, Guibourdenche J, Dionne MD, Le Ray C, Anselem O, Serreau R, Goffinet F, Tsatsaris V. Placental growth factor for the prediction of adverse outcomes in patients with suspected preeclampsia or intrauterine growth restriction. PLoS One. 2012;7(11):e50208. doi: 10.1371/journal.pone.0050208. Epub 2012 Nov 28. PMID 23209675
- [Background] Zeisler H, Llurba E, Chantraine F, Vatish M, Staff AC, Sennstrom M, Olovsson M, Brennecke SP, Stepan H, Allegranza D, Dilba P, Schoedl M, Hund M, Verlohren S. Predictive Value of the sFlt-1:PlGF Ratio in Women with Suspected Preeclampsia. N Engl J Med. 2016 Jan 7;374(1):13-22. doi: 10.1056/NEJMoa1414838. PMID 26735990